CLINICAL TRIAL: NCT05324007
Title: Babies' Expectations About Racial Interactions
Acronym: BEARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Principal Investigator, Hyesung Grace Hwang, Principal Investigator, University of Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB18-1257
Record Dates: First submitted 2022-04-01; First posted 2022-04-12 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Infant Behavior
MeSH Terms: conditions — Infant Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White-White (Experimental): Infants will first view 4 familiarization trials, in which the two adults each take turns waving and saying a short sentence. Each trial will last 10.5s. Which adult speaks first and which side she appears on will be counterbalanced. These familiarization trials will ensure infants encode each person separately. Then infants will watch 6 test trials (3 affiliation and 3 disengagement). The test trials will alternate, and the order will be counterbalanced across infants. In affiliation trials, the two adults will say "hello" and wave, whereas in the disengagement trials, the two adults will say "hmph", and turn away from each other. Both affiliation and disengagement will have the same length (3s), with actors maintaining the same distance from each other throughout the video. The procedure will be identical for all arms except in "White-White" arm, the two adults infants see will be two White adults.
  Interventions: Other: Basic Science
- Black-Black (Experimental): The procedure is identical to the "White-White" arm except the two adults infants see will be two Black adults.
  Interventions: Other: Basic Science
- Black-White (Experimental): The procedure is identical to the "White-White" arm except the two adults infants see will be one White and one Black adult.
  Interventions: Other: Basic Science

INTERVENTIONS:
Other: Basic Science — This is a basic science experiment to test whether infants' looking time to video stimuli differ according to the race of the individuals shown.

SUMMARY:
This study will examine whether infants view race as an inductively useful social cue to predict third-party social relationships.

DETAILED DESCRIPTION:
Based on findings that infants expect more affiliation between same language speakers than different language speakers (i.e., infants will look longer at affiliation between different language speakers than same language speakers), this study will assess whether infants' expectations about intra- and inter-racial interactions will also follow the same pattern as language. After informed consent, participants who meet the eligibility requirements will be randomized into one of the 3 conditions: Watching (1) two White adults affiliating and disengaging, (2) two Black adults affiliating and disengaging, and (3) one White and one Black adults affiliating and disengaging.

ELIGIBILITY:
Inclusion Criteria:

* full term (at least 37 weeks at birth)
* no known developmental delays

Exclusion Criteria:

* not full term (less than 37 weeks at birth)
* known developmental delays

Ages: 8 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyesung G Hwang, PhD, Principal Investigator — University of Chicago
Locations (1):
- Infant Learning and Development Laboratory at University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All data that was used in analysis will be shared publicly on Open Science Framework repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Once data has been collected and cleaned it will be available to the public indefinitely.
Access Criteria: Anonymized individual participant data will be publicly available for anyone to access on Open Science Framework repository.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants were recruited and tested through an online platform called Lookit (lookit.mit.edu), a website developed by MIT researchers to test infants from the comforts of their homes.
Pre-assignment Details: No participants were excluded before assignment to arm.
Period: Overall Study
Arm/Group | White-White | Black-Black | Black-White
Started | 43 | 43 | 42
Completed | 30 | 30 | 30
Not Completed | 13 | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | White-White | Black-Black | Black-White | Total
Number analyzed (Participants) | 43 | 43 | 42 | 128
Age, Continuous [Mean (Standard Deviation); unit: days] — Age in days
  days | 333.09 (72.66) | 336.33 (64.06) | 327.64 (69.89) | 332.39 (68.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 17 | 58
  Male | 21 | 24 | 25 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 6 | 7 | 7 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 28 | 28 | 29 | 85
  More than one race | 7 | 6 | 6 | 19
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 43 | 42 | 128

OUTCOME MEASURES:

1. Primary Outcome: Participants' Average Time Spent Looking at Stimuli According to Condition
Description: Infants' looking time to affiliation vs. disengagement stimuli was measured by two coders blind to the condition that infants were assigned to. Then, the values from each coders were compared and if there was disagreement, after discussion one value was selected. Thus, the reported outcome is the single value that both coders produced or agreed upon values from the two coders.
Time Frame: After the infants completed the study (which lasted about 10 minutes), two coders viewed the video recording of the session to measure infants' looking at the affiliation and disengagement stimuli.
Population: We ended up excluding 38 infants from the 128 infants we recruited due to technical issues (e.g., no video of infant in the study produced or infants' study video was cut off due to internet speed), parental/family interference (e.g., parents spoke during the study or siblings interrupted), and due to infant crying and not completing the study. Thus, after exclusion, the final data sample we analyzed is 90 infants.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | White-White | Black-Black | Black-White
Number analyzed (Participants) | 30 | 30 | 30
seconds
  Avg looking at affiliation | 10.72 (3.27) | 10.07 (3.20) | 10.99 (3.56)
  Avg looking at disengagement | 9.53 (3.10) | 10.20 (2.45) | 9.65 (3.52)
Statistical Analysis 1: Comparison: White-White vs Black-Black vs Black-White; We will examine whether looking time at affiliation will be greater when looking at Black-White interactions than at White-White or Black-Black interactions. That is, we will test if infants will be more surprised (look longer) by affiliation between different-race people interacting than same race people interacting. We will conduct a mixed ANOVA with conditions (Black-White, White-White, Black-Black) as a between-subject and test type (affiliation vs. disengagement) as within-subject factors; Test type: Equivalence — Estimated effect size was based on Liberman et al. (2017) that found a partial eta squared of .478 for the interaction between different-language and same-language conditions. Using G*power using an alpha of .05, our target sample size of 30 per condition should provide 99.73% power to detect the main effect in the White-White and Black-Black condition and 99.99% power to detect the main effect in the Black-White condition; p < .05, ANOVA; partial eta squared = .062

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study
Arm/Group | White-White | Black-Black | Black-White
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT05324007/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT05324007/ICF_001.pdf